CLINICAL TRIAL: NCT01902615
Title: Multicenter, Observational, Retrospective Study to Assess the Therapeutic Effectiveness of a Strategy of Induction With Enfuvirtide Within an Optimized Regimen of Antiretroviral Drugs (ARV) in Patients Infected With HIV-1 in Routine Clinical Practice
Brief Title: An Observational Study of Induction Therapy With Fuzeon (Enfuvirtide) in Combination With Antiretroviral Drugs in Patients With HIV-1 Infection
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25313
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, retrospective, observational study will evaluate the therapeutic effectiveness of a strategy of induction with Fuzeon (enfuvirtide) within an optimized regimen of antiretroviral drugs in patients with HIV-1 infection in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* HIV-1+ infection
* Patients with a viral load > 50 copies/ml who have received induction treatment with Fuzeon in combination with antiretroviral treatment
* Naïve for Fuzeon at initiation of induction treatment
* Antiretroviral treatment of at least 12 months duration

Exclusion Criteria:

* Patients who did not receive Fuzeon treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HIV-1 infection having received induction therapy with Fuzeon and antiretroviral drugs
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2001-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Response rate: Proportion of patients with reduction of viral load to < 50 copies/ml | approximately 24 months

SECONDARY OUTCOMES:
Duration of treatment with Fuzeon | approximately 24 months
Time to undetectability, defined as time from initiation of treatment to first observation of viral load < 50 copies/ml | approximately 24 months
Safety: Incidence of adverse events | approximately 24 months
Treatment regimen: Antiretroviral drugs used | approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Barcelona, Barcelona, Spain